CLINICAL TRIAL: NCT02664662
Title: Effectiveness of Tailored Rehabilitation Education on Health Literacy and Health Status of Postoperative Patients With Breast Cancer: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Medical University Hospital
Record Dates: First submitted 2015-12-27; First posted 2016-01-27 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2016-01

CONDITIONS: Health Behavior
Keywords: Breast cancer; Health literacy; Tailored education; Rehabilitation; International Classification of Functioning, Disability and Health
MeSH Terms: conditions — Health Behavior; Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tailored education (Experimental): Tailored rehabilitated education is which fit for each breast cancer patients after surgery in clinic. We design three of tailored books for experimental group. Each patients will be tailored by three principles. First, the educated times and hours are depended on patients physical function and learning ability. Second, the material is depended on each patient's life experience. Finally, the educated content is depended on patient's operation method.
  Interventions: Other: tailored education
- standard education (No Intervention): Only provide one paper of post operation and give education of rehabilitated exercise

INTERVENTIONS:
Other: tailored education — Tailored rehabilitated education is which fit for each breast cancer patients after surgery in clinic. We design three of tailored books for experimental group. Each patients will be tailored by three principles. First, the educated times and hours are depended on patients physical function and learning ability. Second, the material is depended on each patient's life experience. Finally, the educated content is depended on patient's operation method.
  Arms: tailored education

SUMMARY:
For the past few years, the survival rate of breast cancer improved due to the advancement of surgery techniques and popularization of cancer screening. However, prolonged survival rate is definitely not equal to achieving a sound quality of life among breast cancer survivors. The health status of cancer survivors might deteriorate according to the severe side effect of multiple therapies.

Health literacy is the ability to access, understand, evaluate and communication information as a way to promote and maintain health. Therefore, good health literacy raise the quality of life of breast cancer survivors by a good competence in searching and using medical resources. Moreover, how to improve health literacy after cancer surgery becomes an important part recently. Even if the most fundamental concept has promoted for decades, the clinical workers still use the identical education of medical care after surgery for breast cancer survivors. However, the identical education is not appropriate for each of patients. In fact, each of breast cancer survivors has the different cancer stage leading to accept different therapy and producing different side effect. Besides, the background and the role of life are very different from each other. Because of the above reasons, the aim of the study is going to develop a tailored rehabilitated education, which fit for each breast cancer patients after surgery in clinic. At the same time, the health literacy ability might be improved by tailored rehabilitated education. When health literacy level is raised, the breast cancer survivors have a good quality of life and beautiful health status.

DETAILED DESCRIPTION:
This evaluator-blinded, randomized, prospective, controlled trial enrolled consecutive patients who fulfilled the inclusion criteria. Patients were stratified into four strata according to the side of the lesion and the surgical approach. A set of numbered envelopes containing cards indicating the allocated group was prepared for each stratum. When a new eligible participant was registered, an envelope was randomly drawn, and the therapist was informed of group allocation.

To ensure consistent intervention, two certified occupational therapists were trained by two primary investigators to administer the intervention and control group protocols independently. The two trained occupational therapists recorded outcome measurements at the baseline and immediately after the intervention. The evaluators were blinded to group allocation, and participants were blinded to the study hypotheses.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient has been diagnosed breast cancer (age > 20)
2. Have a good motivation and cooperation when accept breast cancer education
3. Read words or speak in Chinese fluently

Exclusion Criteria:

1. Diagnoses mental problems
2. Patient with Cancer terminal stage and weakness

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Health literacy Assessments in breast cancer | one month
  The Health Literacy scale is five point likert scale of choices, which is evaluated by patient. There are 47 items and the higher scores means the higher literacy performance.

SECONDARY OUTCOMES:
Disability of Arm Shoulder and Hand(DASH) | one month
  DASH evaluate the patient's hand function. There are 15 items and get higher get higher hand function performance
Barthel Index | one month
  Barthel Index is an assessment tool which evaluate activity participated performance. There are 10 items and higher scores means higher activity participated performance.
Frenchay activities index (FAI) | one month
  FAI is an assessment tool which evaluate instrumental activity participated performance. There are 15 items and higher scores means higher performance.
EuroQol-5 dimension (EQ5D) | one month
  EQ5D is an assessment tool which evaluate quality of life. There are 5 items and 1 visual analogue scale. The higher scores means good quality of life performance.
Brief Symptom Rating Scale | one month
  Brief Symptom Rating Scale is an assessment tool which evaluate the psychosis performance. There are 6 items and higher scores means good psychosis performance.

CONTACTS AND LOCATIONS:
Overall Officials: Bi-Chu Lin, Study Director — Taipei Medical University; Wen-Hsuan Hou, Study Director — Taipei Medical University
Locations (1):
- Huang Szu-Chi, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol